CLINICAL TRIAL: NCT02888990
Title: An Open Label Phase II Study to Evaluate the Efficacy and Safety of Induction and Consolidation Therapy With Dasatinib in Combination With Chemotherapy in Patients Aged 55 Years and Over With Philadelphia Chromosome Positive (Ph+ or BCR-ABL+) Acute Lymphoblastic Leukemia (ALL).
Brief Title: Dasatinib and Low Intensity Chemotherapy for Ph+ Acute Lymphoblastic Leukemia
Acronym: EWALLPH01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Philippe ROUSSELOT, study coordinator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-005694-21
Record Dates: First submitted 2016-08-19; First posted 2016-09-05 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-08

CONDITIONS: Leukemia, Lymphoblastic, Acute
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Arm (Experimental): standard treatment + dasatinib
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib

SUMMARY:
1. The use of imatinib in combination or in association with chemotherapy is now considered as the gold standard for the treatment of Ph+ ALL. The complete remission (CR) rate is 90% versus 20% to 40% with chemotherapy alone. The combination of imatinib, vincristine and dexamethasone is a well tolerated regimen in aged patients and is also associated with a high CR rate of 80% to 90% in patient aged 55 years and over.
2. However, despite high CR rates, the progression free survival rate at 12 months of patients treated with the combination of imatinib and chemotherapy is 30% to 50%. Relapses remain frequent and only patients intensified with allogenic haematopoietic stem cell transplantation are in long term remission. This strategy is not fully applicable to most patients aged 55 years and over.
3. Relapses after or during imatinib therapy in patients with Ph+ ALL are associated with BCR-ABL tyrosine kinase domain mutation in 80% of cases, predominantly of the p-loop. The exact incidence of the T315I mutation is controversial and can be estimated to be near 50%. Conversely, the detection of the T315I or F317 mutation in a patient is a very strong predictor of relapse.
4. Dasatinib is a potent SCR and BCR-ABL tyrosine kinase inhibitor with preserved in vitro activity in most of the BCR-ABL mutated cell lines, except for the T315I and F317 mutations. This is also the case in vivo, with patients harbouring BCR-ABL TK domain mutations remaining sensitive to dasatinib. The CHR rate in Ph+ ALL resistant to imatinib is 33% and the median progression-free survival is 3.7 months. Progression free survival (PFS) rate at 12 months is 22%.

The goal of this trial is to evaluate the efficacy and the tolerance of the combination of dasatinib with chemotherapy in the front-line setting as induction and consolidation therapy in Ph+ ALL patient aged 55 years and over. A European consensus has been reached to adopt a common chemotherapeutic schedule for patients aged 55 years and over. This schedule will be used in this trial with the addition of dasatinib as concomitant therapy during induction and alternating with chemotherapy during consolidation and maintenance. A CR rate of 90% and a progression free survival of 60% at 12 months are expected. The patients will be prospectively monitored for minimal residual disease and mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 55 years
2. Philadelphia chromosome or BCR-ABL positive acute lymphoblastic leukaemia
3. Not previously treated except with corticosteroids or single dose vincristine (three doses cyclophosphamide accepted but not recommended)
4. With or without documented CNS involvement
5. Signed written inform consent
6. Molecular evaluation for BCR-ABL done

Exclusion Criteria:

1. Patients with ECOG status > 2
2. Patient previously treated with Tyrosine Kinase Inhibitors
3. Patients with QTc > 470 ms
4. Heart insufficiency NYHA grade III/IV, LEVF < 50% and or RF < 30%, myocardial infarction within the past 6 months prior to study
5. Active secondary malignancy
6. Patients with active bacterial, viral or fungal infection
7. Known infection with HIV, Hepatitis B (except post vaccinal profile) or C
8. Treatment with any, other investigational agent or participating in another trial within 30 days prior to entering this study
9. Inadequate hepatic functions defined as ASAT or ALAT > 2,5 times the institutional upper limit of normal and total bilirubin > 2 fold the institutional upper limit unless considered to be due to organ involvement by the leukemia
10. Concurrent severe diseases which exclude the administration of therapy

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-08; Primary Completion 2011-05 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival at 12 months | 12 months

SECONDARY OUTCOMES:
The proportion of Complete haematological remission | 5 years
The proportion of Major molecular response defined by a BCR-ABL/ABL ≤ 0.1% in bone marrow | 5 years
The proportion of Complete molecular response | 5 years
Event free survival | 5 years
Relapse free survival | 5 years
Progression free survival | 5 years
The proportion of Detection of a T315I or F317 BCR-ABL TK mutation | 5 years
The proportion of Molecular progression | 5 years
Overall survival | 5 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years
Death during induction | 2 months
Death in complete remission | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rousselot Philippe, MD, Principal Investigator — CH Versailles
Locations (64):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU Ambroise Paré, Mons
- France (57):
  - Centre Hospitalier Départemental FELIX GUYON, Saint-Denis, La Reunion
  - Ch D'Aix En Provence, Aix-en-Provence
  - Groupe Hospitalier Sud, Amiens
  - CHU Angers, Angers
  - Chr Annecienne, Annecy
  - Ch Victor Dupouy, Argenteuil
  - CHG D'Avignon Henri Duffaut, Avignon
  - C.H. de la Côte Basque, Bayonne
  - Hôpital JEAN MINJOZ, Besançon
  - CH Blois, Blois
  - Avicenne, Bobigny
  - CHU Brest, Brest
  - Hôpital CLEMENCEAU, Caen
  - HIA Percy, Clamart
  - Hotel Dieu, Clermont-Ferrand
  - Hôpital PASTEUR, Colmar
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Henry Mondor, Créteil
  - Hôpital du BOCAGE, Dijon
  - CH Dunkerque, Dunkirk
  - Hôpital A. MICHALLON, Grenoble
  - CH Versailles, Le Chesnay
  - CH Lens, Lens
  - Hopital Claude Huriez, Lille
  - Hôpital Dupuytren, Limoges
  - Edouard Herriot, Lyon
  - IPC, Marseille
  - CH Meaux, Meaux
  - Hôpital Notre Dame de Bon Secours, Metz
  - Hôpital LAPEYRONIE, Montpellier
  - CH E Muller, Mulhouse
  - Hotel Dieu, Nantes
  - Archet 1, Nice
  - CHU Nimes, Nîmes
  - Hôpital de la Source, Orléans
  - Cochin, Paris
  - Hopital St louis, Paris
  - Necker, Paris
  - Pitie Salpetrière, Paris
  - St Antoine, Paris
  - CH Perpignan, Perpignan
  - Hôpital du HAUT LEVEQUE, Pessac
  - Hopital Lyon Sud, Pierre-Bénite
  - CHU Mileterie, Poitiers
  - Hopital R Debre, Reims
  - Hôpital de PONTCHAILLOU, Rennes
  - CH Victor PROVO, Roubaix
  - Centre HENRI BECQUEREL, Rouen
  - centre rene Huguenin, Saint-Cloud
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - CHU Hautepierre, Strasbourg
  - HIA Ste Anne, Toulon
  - Hôpital de PURPAN, Toulouse
  - CHU Tours, Tours
  - Hotel Dieu, Valenciennes
  - CH Brabois, Vandœuvre-lès-Nancy
  - IGR, Villejuif
- Germany (2):
  - St. Johannes-Hospital, Duisburg
  - Robert Bosch-Krankenhaus, Stuttgart
- Italy (3):
  - Ospedali Riuniti di Bergamo, Bergamo
  - Ospedale San Gerardo, Monza
  - Dipartimento Oncologico La Maddalena, Palermo

IPD SHARING:
Plan to Share IPD: No